CLINICAL TRIAL: NCT04425395
Title: The Effect of Nonverbal Vocalisations on Pain Tolerance
Acronym: VOCPAIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Laboratoire ENES-CNPS (Université Lyon/Saint Etienne) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 19CH216; 2020-A00277-32 (Other: ANSM)
Record Dates: First submitted 2020-06-08; First posted 2020-06-11 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Healthy
Keywords: nonverbal vocal communication; pain tolerance; cold pressor test; Nociception Level Index; Video pupillometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy adult population aged 18 to 60 years. (Experimental): Their pain tolerance will be tested using the Cold Pressor Task while producing vocalisations. Produced vocalisations will be audio recorded and physiological measures will be taken using two techniques: Nociception Level Index and video pupillometry.
  Interventions: Behavioral: Cold pressor task (CPT); Behavioral: Acoustic Recordings; Diagnostic Test: Index measurement NOL™; Diagnostic Test: Video pupillometry

INTERVENTIONS:
Behavioral: Cold pressor task (CPT) — The cold pressor test is among the most common and established methods for studying human reactions to pain and pain tolerance. Participants submerge a hand in cold water (approx. 5°C) and are asked to keep their hand submerged for as long as can (until the sensation is intolerable), up to a maximum of 5 min. The procedure is safe because the hand is removed before adverse effects can occur. The participant will be given a break of 5 min in between trials, and will interchange hands between trials. During this break hand may to be place in warm water (25-35°C) for up to 4 min to normalise hand temperature, which will be measured before and after each trial using a digital thermometer held firmly in the palm of the hand.
  Each participant will complete no more than three trials (conditions) in a randomised order.
Behavioral: Acoustic Recordings — During the experiment, the vocalizations produced will be systematically recorded for each participant and an analysis of the acoustic structure of these vocalizations will be carried out.
Diagnostic Test: Index measurement NOL™ — Four sensors placed non-invasively on one finger. of the participants will be able to calculate a dozen physiological parameters converts in real time into a pain index called NOL (for Nociception Level Index).
Diagnostic Test: Video pupillometry — This technique is based on the observation of the dilatation of the pupil during the perception of a nociceptive stimulus in test persons.

SUMMARY:
Humans produce non-verbal vocalizations (shouting, growling, screaming), laughter, ...) in various contexts that are likely to perform biological functions.

and important social issues. Yet despite their importance in the human vocal repertoire, the mechanisms and functions of non-verbal vocalizations remain little studied and poorly understood including in humans. In this context, the investigators wish to examine how the production of vocalizations non-verbal communication influences pain tolerance in healthy adults.

DETAILED DESCRIPTION:
Humans produce nonverbal vocalisations such as screams, grunts, roars, cries and laughter across a variety of contexts. Yet despite the prominence and apparent importance of these nonverbal sounds in human communication, the investigators still know very little about their influence on human perception and behaviour. That's why, in this study, the investigators will examine specifically the influence of nonverbal vocal production on pain tolerance.

The remainder of the study will involve up to three trials of a pain tolerance (cold pressor) task, during which the investigators will ask participants to produce vocalisations (e.g., screams or words) while submerging the participant's hand in bath of circulating cold water.

The results of the study will contribute to our theoretical understanding of the functions of nonverbal vocal communication in humans, in particular the influence of nonverbal vocal production (i.e., yelling) on pain tolerance.

ELIGIBILITY:
Inclusion Criteria:

* Participant in good health
* Affiliated or entitled participant in a social security scheme
* Participant who has received informed information about the study and has co-signed a consent to participate in the study with the investigator.

Exclusion Criteria:

* Chronic pain
* High blood pressure or poor circulation
* Cardiac or vascular disease, or a heart condition (including symptoms of Raynaud's syndrome)
* Allergy or hypersensitivity to cold
* Diabetes
* Epilepsy
* Pregnancy
* Recent serious injury
* Neurological or psychiatric condition known to affect pain tolerance (e.g., peripheral neuropathy, schizophrenia)
* History of fainting or seizures
* History of frostbite
* Chronic smoker (more than 10 cigarettes a day)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Estimated)
Dates: Start 2022-05-11 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Pain tolerance | at inclusion
  Delay (in seconds) in removing the hand when testing the Cold Pressor.

SECONDARY OUTCOMES:
Onset of pain | at inclusion
  Participant verbally indicates when he or she begins to feel the sensation of pain (time of onset measured in seconds)
Pain intensity | at inclusion
  Subjective assessment of maximum pain intensity by participants for a given trial.
  Measured by scale of 0 (no pain) at 100 (extreme pain).
correlation between NOL index and pupillary diameter | at inclusion
  Measurement of the NOL index (index ranging from 0 to 100) and measurement of pupillary diameter (in mm) and its variations in response to nociceptive stimuli by video pupillometry.
Analysis of Acoustic Recordings | at inclusion
  Using a dedicated script in software specialised in acoustic analysis (e.g. PRAAT).

CONTACTS AND LOCATIONS:
Overall Officials: Roland PEYRON, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Centre Hospitalier Universitaire Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No